CLINICAL TRIAL: NCT00626535
Title: A Multicenter, Randomized, Double-Blind Parallel-Group, Placebo-Controlled Efficacy Study Comparing 4 Weeks of Treatment With Esomeprazole 20 mg Once Daily to Placebo qd for the Resolution of Upper Abdominal Pain in Patients With Symptomatic Gastroesophageal Reflux Disease (sGERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9619C00001
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Symptomatic Gastroesophageal Reflux Disease (sGERD)
Keywords: Symptomatic Gastroesophageal Reflux Disease (sGERD); Nexium; Esomeprazole
MeSH Terms: interventions — Esomeprazole

ARMS (2):
- 1 (Experimental): 20mg once daily
  Interventions: Drug: Esomeprazole
- 2 (Placebo Comparator): Oral once daily
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Esomeprazole — 20mg Oral Once Daily
  Other Names: Nexium
  Arms: 1
Drug: Matching placebo — Oral Once Daily
  Arms: 2

SUMMARY:
This study compares 4 weeks of treatment with Esomeprazole 20 mg once daily to Placebo in the treatment of Upper Abdominal Pain in patients with Symptomatic Gastroesophageal Reflux Disease (sGERD)

ELIGIBILITY:
Inclusion Criteria:

* History of episodes of heartburn and upper abdominal pain for 6 months or longer.
* Episodes of heartburn 2 or more days during the 7 days prior to the screening visit. Moderate or severe upper abdominal pain on at least 3 out of the 7 consecutive days of the run-in period.
* A normal endoscopy within 14 days of Visit 1 of between Run-in and randomization.

Exclusion Criteria:

* Subjects with pain likely to be due to irritable bowel syndrome (IBS)
* History of esophageal, gastric or duodenal surgery, except for closure of an ulcer.
* History of severe liver disease, including (but not limited to) cirrhosis and acute or chronic hepatitis.
* Further diseases / conditions, as listed in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2003-03; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
To demonstrate a difference between esomeprazole 20 mg once daily and placebo qd in the resolution and relief of upper abdominal pain after 4 weeks of treatment in patients with sGERD | Daily diary cards completed by the patient

SECONDARY OUTCOMES:
To demonstrate a difference between esomeprazole 20 mg once daily and placebo qd in the resolution and relief of upper abdominal pain after 1, 2, and 4 weeks of treatment in patients with sGERD | Daily diary cards completed by the patient
To demonstrate a difference in percentage of days with, days to resolution of, and severity of upper abdominal pain through 4 weeks of treatment between esomeprazole 20 mg once daily and placebo qd in patients with sGERD | Percentage of days without upper abdominal pain over the 4-week treatment period
To assess the safety and tolerability of esomeprazole 20 mg qd through 4 weeks of treatment. | Mean severity of the patient's upper abdominal pain over the last 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca